CLINICAL TRIAL: NCT00632359
Title: A Study of Lenalidomide in Patients With Chronic Lymphocytic Leukemia and Residual Disease After Chemotherapy - RV-CLL-PI-0270
Brief Title: Lenalidomide in Chronic Lymphocytic Leukemia (CLL) Patients With Residual Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0213; NCI-2012-01690 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2008-03-03; First posted 2008-03-10 (Estimated); Results first posted 2020-02-10 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-01

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Chronic Lymphocytic Leukemia; CLL; Lenalidomide; Revlimid
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lenalidomide (Experimental): Lenalidomide 10 mg daily given for 12 months.
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — 10 mg daily given for 12 months
  Other Names: Revlimid

SUMMARY:
The goal of this clinical research study is to learn if Revlimid (lenalidomide) can help to reduce the level of leukemia in your body. The safety of this drug will also be studied.

DETAILED DESCRIPTION:
The Study Drug:

Lenalidomide is designed to change the body's immune system and may also interfere with the development of tiny blood vessels that help support tumor growth. Therefore, in theory, it may decrease or prevent the growth of cancer cells.

Study Drug Administration:

If you are found to be eligible to take part in this study, you will take lenalidomide by mouth every night each day for up to 12 months. You should swallow lenalidomide capsules whole, with water, at the same time each day. Do not break, chew, or open the capsules. If you miss a dose of lenalidomide, take it as soon as you remember on the same day. If you miss a dose, it should not be made up on another day.

The dose and schedule of lenalidomide may be changed, depending on the side effects you may experience.

Study Visits:

Once a week during the first 4 weeks, blood (about 1 tablespoon) will be drawn for routine tests. Blood may be drawn more often if the dose of lenalidomide needs to be changed or if you experience side effects.

After the first 4 weeks, blood (about 1 tablespoon) will be drawn for routine tests every 2 weeks until the doctor thinks your dose of lenalidomide will not change. After this, blood (about 1 tablespoon) will then be drawn every 4 weeks for routine tests.

On Month 4 and 12 (+14 days), you will have a physical exam and blood (about 2-3 teaspoons) will be drawn to check the status of the disease.

On Month 4 and 12 (+14 days), and then every 3 months after that (unless your study doctor does not think it is necessary), you will have a bone marrow biopsy and aspirate to check the status of the disease.

Length of Study:

You will continue receiving the study drug for up to 12 months. You will continue having study visits for as long as the disease remains stable. You will be taken off study early if the disease gets worse or intolerable side effects occur.

ELIGIBILITY:
Inclusion Criteria:

1. Patients should have completed their chemotherapy 3 months prior to start of treatment with lenalidomide and not more than 9 months prior to treatment initiation.
2. Patients with CLL/Small Lymphocytic Lymphoma (SLL) that achieve a complete or stable partial remission after combination of chemotherapy. Patients in complete remission need to have documentation of residual disease by immunophenotyping and/or PCR molecular testing.
3. Eastern Cooperative Oncology Group (ECOG)/World Health Organization (WHO) status of 0-2.
4. Adequate renal and hepatic function (creatinine equal to or less than 2mg/dL - total bilirubin equal to or less than 2).
5. Females of childbearing potential (FCBP). A female of childbearing potential is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; 2) or has not been naturally postmenopausal for at least 24 consecutive months (has NOT had menses at any time in the preceding 24 consecutive months).
6. FCBP must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10-14 days prior to and again within 24 hours of starting lenalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control; one highly effective and one additional effective method AT THE SAME TIME at least 28 days before starting taking lenalidomide.
7. FCBP must also agree to ongoing pregnancy testing weekly for the first four weeks and then every 28 days while on therapy and at discontinuation of treatment.
8. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy. All patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure.
9. Age 18 and older.
10. Signed, written IRB-approved informed consent.

Exclusion Criteria:

1. Known sensitivity to lenalidomide or thalidomide or it's derivatives
2. Known positivity for HIV or active hepatitis B or C.
3. Pregnant or breast feeding females. Lactating females must agree not to breast feed while taking lenalidomide.
4. History of tuberculosis within the last five years or recent exposure to tuberculosis equal to or less than 6 months.
5. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
6. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
7. Use of any other experimental drug or therapy within 28 days of baseline.
8. Concurrent use of other anti-cancer agents or treatments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2008-02; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Ferrajoli, M.D,, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: February 28, 2008 to January 7, 2015. All recruitment done at The University of Texas MD Anderson Cancer Center.
Period: Overall Study
Arm/Group | Lenalidomide
Started | 33
Completed | 31
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Lenalidomide
Number analyzed (Participants) | 33
Age, Continuous [Median (Full Range); unit: years] | 59 [39 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 32
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Quality of Remission: Number of Participants With Response Versus No Response by NCI Working Group Criteria Disease Status Change at Start/End of Lenalidomide Consolidation
Description: To evaluate ability of lenalidomide to improve quality of remission (e.g. from partial remission (PR) to complete remission (CR)), disease status assessed at start & end of Lenalidomide consolidation. NCI Working Group Response Criteria: Participants who began therapy in PR, improvement of status to nodular partial remission (nPR) or CR; Participants in nPR (otherwise CR, bone marrow nodules identified histologically), improvement of status to CR. Participants in CR, resolution of measurable disease in blood &/or bone marrow per immuno flow cytometry or PCR testing. Progressive Disease (PD): One or more of following: >50% increase in sum of products of =/>2 lymph nodes on 2 consecutive examinations; One+ node must be >2 cm or appearance of new enlarged lymph nodes; >50% increase in liver &/or spleen as determined by physical examination/appearance of splenomegaly not previously present; >50% increase in circulating lymphocytes with absolute count >10,000.
Time Frame: Baseline to 12 Months, Disease status assessed at Start/End of Lenalidomide Consolidation
Population: Of the three participants registered, two were not evaluable for response.
Measure: Number; unit: participants
Arm/Group | Lenalidomide
Number analyzed (Participants) | 31
participants
  Response | 10
  No Response | 21

2. Primary Outcome: Response Assessments: Disease Status at the End of Lenalidomide Consolidation Per International Workshop on Chronic Lymphocytic Leukemia (IWCLL) Response Criteria
Description: Complete remission (CR), requiring absence of peripheral blood clonal lymphocytes by immunophenotyping, absence of lymphadenopathy, absence of hepatomegaly or splenomegaly, absence of constitutional symptoms and satisfactory blood counts; positive or negative minimal residual disease (MRD); Partial remission (PR), defined as ≥ 50% fall in lymphocyte count, ≥ 50% reduction in lymphadenopathy or ≥ 50% reduction in liver or spleen, together with improvement in peripheral blood counts; Nodular Partial Remission (nPR) is CR with bone marrow nodules identified histologically. Progressive disease (PD), defined as ≥ 50% rise in lymphocyte count to > 5 x109/L, ≥ 50% increase in lymphadenopathy, ≥ 50% increase in liver or spleen size, Richter's transformation, or new cytopenias due to CLL; Stable disease, defined as not meeting criteria for CR, PR or PD.
Time Frame: 12 Months, Disease status assessed at the End of Lenalidomide Consolidation
Population: Of the 33 participants who were treated, two Participants were not evaluable.
Measure: Number; unit: participants
Groups:
- Assessment at End of Consolidation: Response following 12 months of Lenalidomide 10 mg daily.
Arm/Group | Assessment at End of Consolidation
Number analyzed (Participants) | 31
participants
  CR, MRD Positive or Negative | 13
  PR | 8
  nPR | 7
  PD | 1

3. Primary Outcome: Time to Progression
Description: Time from the start of study drug therapy to the first documentation of disease progression. Progressive disease characterized by at least one of the following: >50% increase in the sum of products of at least 2 lymph nodes on 2 consecutive examinations. At least one node larger than 2 cm. Or, appearance of new enlarged lymph nodes. >50% increase in size of liver and/or spleen as determined by physical examination or appearance of splenomegaly which was not previously present. >50% increase in number of circulating lymphocytes with absolute count of at least 10,000.
Time Frame: From baseline to 12 months
Population: Of the 33 participants treated, two were not evaluable for outcome assessment due to early departure from study.
Measure: Mean (95% Confidence Interval); unit: Months
Arm/Group | Lenalidomide
Number analyzed (Participants) | 31
Months | 8 [6.6 to 9.4]

ADVERSE EVENTS:
Time Frame: Adverse event collection for 12 months of treatment.
Arm/Group | Lenalidomide
Serious Adverse Events (participants affected / at risk) | 8/33
Other Adverse Events (participants affected / at risk) | 27/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide (N=33)
Neutropenia (Blood and lymphatic system disorders) | 8 (8)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) — THROMBOSIS/THROMBUS/EMBOLISM
Pulmonary Embolus (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infections, Respiratory syncytial virus (RSV) (Infections and infestations) | 1 (1)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
THROMBOSIS/THROMBUS/EMBOLISM (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide (N=33)
ALKALINE PHOSPHATASE INCREASE (Investigations) | 1 (2)
ALLERGIC RHINITIS (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Alanine aminotransferase Increased (ALT, SGPT) (Investigations) | 2 (7)
ANOREXIA (Metabolism and nutrition disorders) | 1 (1)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1)
Aspartate aminotransferase increased (AST, SGOT) (Investigations) | 2 (5)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1)
AUDITORY/EAR (OTHER) (Ear and labyrinth disorders) | 1 (1)
BILIRUBIN INCREASED (Blood and lymphatic system disorders) | 1 (1)
CARDIAC ISCHEMIA/INFARCTION (Cardiac disorders) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 6 (6)
COUGH (Respiratory, thoracic and mediastinal disorders) | 8 (8)
CREATININE INCREASED (Investigations) | 6 (8)
DERMATOLOGY/SKIN (OTHER) (Skin and subcutaneous tissue disorders) | 1 (1)
DIABETES (Hyperglycemia) (Metabolism and nutrition disorders) | 1 (1)
DIARRHEA (Gastrointestinal disorders) | 9 (11)
DISTENSION/BLOATING (General disorders) | 3 (3)
DIZZINESS (Nervous system disorders) | 1 (1)
DRY SKIN (Skin and subcutaneous tissue disorders) | 1 (1)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 2 (2)
ENDOCRINE (OTHER: adrenal difference) (Endocrine disorders) | 2 (2)
ERYTHEMA MULTIFORME (Skin and subcutaneous tissue disorders) | 1 (1)
FATIGUE (General disorders) | 16 (17)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 2 (2)
FLATULENCE (Gastrointestinal disorders) | 1 (1)
FLU-LIKE SYNDROME (General disorders) | 2 (2)
GASTRITIS (Gastrointestinal disorders) | 2 (2)
GASTROINTESTINAL (OTHER) (Gastrointestinal disorders) | 1 (1)
HEARING CHANGE (WITHOUT MONITORING) (Ear and labyrinth disorders) | 1 (1)
HEMOGLOBIN INCREASED (Investigations) | 18 (22)
HEMORRHAGE, Genitourinary (Renal and urinary disorders) | 1 (1)
HEMORRHAGE, PULMONARY (NOSE) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
HOT FLASHES (Reproductive system and breast disorders) | 1 (1)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 4 (6)
HYPERNATREMIA (Metabolism and nutrition disorders) | 1 (1)
HYPERTENSION (Metabolism and nutrition disorders) | 2 (2)
HYPERURICEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 1 (2)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 2 (3)
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPONATREMIA (Metabolism and nutrition disorders) | 1 (1)
INFECTION (Infections and infestations) | 2 (2)
INSOMNIA (Psychiatric disorders) | 3 (3)
Leukocytosis (Blood and lymphatic system disorders) | 13 (16)
MAGNESIUM, SERUM-HIGH (Metabolism and nutrition disorders) | 1 (1)
METABOLIC/LABORATORY (OTHER) (Metabolism and nutrition disorders) | 10 (16)
MOOD ALTERATION (AGITATION) (Psychiatric disorders) | 1 (1)
MOOD ALTERATION (ANXIETY) (Psychiatric disorders) | 1 (1)
MOOD ALTERATION (DEPRESSION) (Psychiatric disorders) | 1 (1)
MOTOR SKILLS, AFFECTED (Musculoskeletal and connective tissue disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 5 (5)
NEUROPATHY: SENSORY (Nervous system disorders) | 2 (2)
Neutrophils, AGC (absolute granulocyte counts) Increased (Blood and lymphatic system disorders) | 17 (31)
OBSTRUCTION, GU (BLADDER) (Renal and urinary disorders) | 1 (1)
OCULAR/VISUAL (OTHER) (Eye disorders) | 1 (1)
PHLEBITIS (Infections and infestations) | 1 (1)
Platelet count decreased (Investigations) | 12 (16)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 2 (3)
PULMONARY (OTHER) (Respiratory, thoracic and mediastinal disorders) | 3 (3)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RASH/DESQUAMATION (Skin and subcutaneous tissue disorders) | 8 (11)
RENAL FAILURE (Renal and urinary disorders) | 1 (1)
RENAL/GENITOURINARY (OTHER) (Renal and urinary disorders) | 1 (1)
RESPIRATORY SYMPTOMS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RIGORS/CHILLS (General disorders) | 1 (1)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 (1)
SWEATING (Skin and subcutaneous tissue disorders) | 2 (3)
THROMBOSIS/THROMBUS/EMBOLISM (Vascular disorders) | 1 (1)
TINNITUS (Ear and labyrinth disorders) | 1 (1)
TUMOR FLARE REACTION (Investigations) | 4 (4)
VOICE CHANGES (Nervous system disorders) | 1 (1)
PAIN (General disorders) | 8 (8)
FEVER (General disorders) | 1 (1)
INFECTION (Infections and infestations) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes